CLINICAL TRIAL: NCT04377464
Title: COVID-19 - Quality of Life After Infection
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Joseph Walline, Assistant Professor, Chinese University of Hong Kong
Other Study IDs: NTEC-2020-0227
Record Dates: First submitted 2020-05-04; First posted 2020-05-06 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: COVID-19; Quality of Life
Keywords: COVID-19; Quality of Life; Follow-up
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 Survivors: Patients following-up at the PWH outpatient clinics will be enrolled for further evaluation via telephone follow-up at one, three, and six months after hospital discharge. SF12, EQ-5D-5L and work status standardized quantitative assessments of quality of life will be implemented via telephone follow-up at these time-points.
  Interventions: Other: SF12, EQ-5D-5L and work status standardized quantitative assessments

INTERVENTIONS:
Other: SF12, EQ-5D-5L and work status standardized quantitative assessments — Quality of life assessments

SUMMARY:
This study aims to investigate the quality of life of COVID-19 patients after recovery and discharge from the hospital. Patients following-up at the PWH outpatient clinics will be enrolled for further evaluation via telephone follow-up at one, three, and six months after hospital discharge. SF12, EQ-5D-5L and work status standardized quantitative assessments of quality of life will be implemented via telephone follow-up at these time-points. Previous studies of patients infected with SARS-CoV-1 in 2003 at PWH showed that significant numbers of recovering patients had impaired long-term health status. It is important to see if these same problems also afflict patients infected with the SARS-CoV-2 virus (the novel coronavirus which causes COVID-19).

DETAILED DESCRIPTION:
Nearly two million cases have been documented, and thousands have died of the 2019 coronavirus disease (COVID-19). Hong Kong has seen nearly 1,000 documented cases of COVID-19 as of April 11, 2020. Potentially many more cases have gone unreported. The virus that causes the COVID-19 disease, SARS-CoV2, is a coronavirus, from the same group of viruses as the SARS virus from 2003. Worldwide, COVID-19 has killed many more patients than SARS, yet the two viruses share a similar background.

As the peak of viral infections begins to recede, however, the main priority will shift to the process of recovery. Over the past 17 years, Professor David SC HUI has published multiple follow-up examinations of SARS patients conducted at the Prince of Wales Hospital (PWH) outpatient clinics. He found that SARS patients suffered serious long-term effects after ostensibly recovering from their illnesses. Moreover, healthcare workers, who were disproportionately affected by SARS infections in 2003 were also disproportionately affected by long-term disability. Like SARS, many COVID-19 patients require intensive care, intubation, and aggressive medical therapy. One of the treatments tried for SARS patients was high-dose corticosteroids, which has been associated with avascular necrosis of major joints and long term disability. As the COVID-19 pandemic only started a few months ago, it is still unknown if COVID-19 patients will suffer the same fate as SARS survivors.

Recent COVID-19 research has logically focused on the acute diagnosis and treatment of affected patients in order to avoid short -term morbidity and mortality. Past research looking at SARS outcomes showed that both the six month exercise capacity and health status of SARS survivors was lower than that of normal controls. Sepsis patients also experience serious disease caused by infection, and long-term reductions in quality of life have been described in survivors of sepsis. Patients who survive intensive care go on to show deficits in verbal learning and memory, resulting in limitations in returning to work or school. Many SARS survivors developed post-traumatic stress disorder and other debilitating psychological illnesses. Based on the Hong Kong experience with SARS, the investigators are concerned that COVID-19 survivors are at risk for similar challenges in quality of life after discharge from acute care.

The Accident and Emergency Medicine Academic Unit of the Chinese University of Hong Kong based at PWH has worked on multiple studies involving quality of life. In particular, the investigators have previously collaborated with Professor Hui and the CUHK Department of Medicine and Therapeutics (M&T) on a quality of life follow-up study on SARS patients. As for studying health related quality of life, the investigators currently have an ongoing project examining the subject in trauma patients after discharge.

Several instruments have been widely used in quality of life research, including the 36-Item Short Form Health Survey (SF-36), the 12-Item Short Form Health Survey (SF-12), the World Health Organization Quality of Life Instruments (WHOQOL-BREF), EuroQoL-5D (EQ-5D-5L) and the Short-Form Six-Dimension (SF-6D). Our team has experience using the SF-36, SF-12v2(HK) and the EQ-5D-5L survey instruments for monitoring quality of life in research subjects in Hong Kong. For example, the investigators found that trauma patients in Hong Kong scored significantly worse on the SF-36 twelve months after injury. The investigators also found the most dramatic improvements happened in the first one to six months post-injury, and that 45% of subjects had achieved an excellent outcome by four years post-injury. The SF-12v2(HK) with four week recall is a modified version of the SF-36 to be shorter and quicker to use, while also already translated and validated in Hong Kong. The investigators aim to combine our experience with conducting quantitative quality of life studies with the CUHK Department of M&T's expertise in coronavirus treatment and followup to explore the quality of life of COVID-19 patients in recovery.

The reported mortality rates for COVID-19 has so far been lower than SARS, although the higher absolute numbers of COVID-19 patients mean worldwide deaths are overall much higher. Trauma, sepsis and SARS survivors have all experienced significant long-term morbidity and decreased quality of life as a result of their injuries or infections. A previous study of patients infected with SARS-CoV-1 in 2003 at PWH showed that significant numbers of recovering patients had impaired long-term health status. The question this study hopes to answer is to what degree do COVID-19 patients suffer a similar fate? Has the knowledge gained from the SARS experience led to improved quality of life outcomes compared to SARS survivors? Or do the similarities between the viruses that cause SARS and COVID-19 extend to a reduced quality of life after recovery as well?

ELIGIBILITY:
Inclusion Criteria:

* All adult patients aged ≥18 years who present to the infectious disease follow-up clinic at PWH will be screened for inclusion in this study. The inclusion criteria are age ≥18 years, laboratory-confirmed COVID-19 infection with SARS-CoV-2, and patients who agree to follow-up for up to six months following their first interview.

Exclusion Criteria:

* Patients aged below 18 years will be excluded.
* Patients will be excluded if they meet ANY of the following criteria:
* Patients or their next of kin are unable to communicate in Chinese or English,
* Unwilling or unable to provide written informed consent,
* or Patients who will not be available for telephone follow-up at the scheduled times.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: As of April 10, 2020, in the NTEC Hospital Authority cluster there have been 89 patients admitted to PWH (of which 17 patients have already been discharged) and 117 admitted to United Christian Hospital with 42 discharged so far.22 Both PWH and United Christian Hospital's COVID-19 patients will follow-up at the PWH infectious diseases specialist outpatient follow-up clinic. Based on prior studies at PWH with SARS patients, approximately 80% agreed to participate in follow-up studies, so we will likely enroll approximately 200 COVID-19 patients.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-05-05 (Estimated); Primary Completion 2021-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Six-month SF-12v2(HK) Scores | July 1, 2020-January 31, 2021
  The primary outcome measure will be the health summary scores from Short Form Health Survey version 2 Hong Kong (SF-12v2(HK)) in COVID patients at six-months post-discharge from hospital.

SECONDARY OUTCOMES:
Six-month EQ-5D-5L Scores | July 1, 2020-January 31, 2021
  The secondary outcome measures will include the health status measures of the EuroQuality of Life Five Dimensions (EQ-5D-5L) at six-months.
One-month SF-12v2(HK) | July 1, 2020-January 31, 2021
  The secondary outcome measures will include the health status measures of the Short Form Health Survey version 2 Hong Kong (SF-12v2(HK)) at one-month.
One-month EQ-5D-5L Scores | July 1, 2020-January 31, 2021
  The secondary outcome measures will include the health status measures of the EuroQuality of Life Five Dimensions (EQ-5D-5L) at one-month.
Three-month SF-12v2(HK) Scores | July 1, 2020-January 31, 2021
  The secondary outcome measures will include the health status measures of the Short Form Health Survey version 2 Hong Kong (SF-12v2(HK)) at three-months.
Three-month EQ-5D-5L Scores | July 1, 2020-January 31, 2021
  The secondary outcome measures will include the health status measures of the EuroQuality of Life Five Dimensions (EQ-5D-5L) at three-months.
One, Three and Six-month Return to Work Status | July 1, 2020-January 31, 2021
  Return to work status in COVID patients at one, three and six-months post discharge from hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Walline, MD, Principal Investigator — Chinese University of Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhao S, Musa SS, Lin Q, Ran J, Yang G, Wang W, Lou Y, Yang L, Gao D, He D, Wang MH. Estimating the Unreported Number of Novel Coronavirus (2019-nCoV) Cases in China in the First Half of January 2020: A Data-Driven Modelling Analysis of the Early Outbreak. J Clin Med. 2020 Feb 1;9(2):388. doi: 10.3390/jcm9020388. PMID 32024089
- [Background] Li TS, Gomersall CD, Joynt GM, Chan DP, Leung P, Hui DS. Long-term outcome of acute respiratory distress syndrome caused by severe acute respiratory syndrome (SARS): an observational study. Crit Care Resusc. 2006 Dec;8(4):302-8. PMID 17227266
- [Background] Hui DS. Severe acute respiratory syndrome (SARS): lessons learnt in Hong Kong. J Thorac Dis. 2013 Aug;5 Suppl 2(Suppl 2):S122-6. doi: 10.3978/j.issn.2072-1439.2013.06.18. PMID 23977432
- [Background] Bhatraju PK, Ghassemieh BJ, Nichols M, Kim R, Jerome KR, Nalla AK, Greninger AL, Pipavath S, Wurfel MM, Evans L, Kritek PA, West TE, Luks A, Gerbino A, Dale CR, Goldman JD, O'Mahony S, Mikacenic C. Covid-19 in Critically Ill Patients in the Seattle Region - Case Series. N Engl J Med. 2020 May 21;382(21):2012-2022. doi: 10.1056/NEJMoa2004500. Epub 2020 Mar 30. PMID 32227758
- [Background] Griffith JF, Antonio GE, Kumta SM, Hui DS, Wong JK, Joynt GM, Wu AK, Cheung AY, Chiu KH, Chan KM, Leung PC, Ahuja AT. Osteonecrosis of hip and knee in patients with severe acute respiratory syndrome treated with steroids. Radiology. 2005 Apr;235(1):168-75. doi: 10.1148/radiol.2351040100. Epub 2005 Feb 9. PMID 15703312
- [Background] Li Y, Xia L. Coronavirus Disease 2019 (COVID-19): Role of Chest CT in Diagnosis and Management. AJR Am J Roentgenol. 2020 Jun;214(6):1280-1286. doi: 10.2214/AJR.20.22954. Epub 2020 Mar 4. PMID 32130038
- [Background] Shanmugaraj B, Siriwattananon K, Wangkanont K, Phoolcharoen W. Perspectives on monoclonal antibody therapy as potential therapeutic intervention for Coronavirus disease-19 (COVID-19). Asian Pac J Allergy Immunol. 2020 Mar;38(1):10-18. doi: 10.12932/AP-200220-0773. PMID 32134278
- [Background] Gautret P, Lagier JC, Parola P, Hoang VT, Meddeb L, Mailhe M, Doudier B, Courjon J, Giordanengo V, Vieira VE, Tissot Dupont H, Honore S, Colson P, Chabriere E, La Scola B, Rolain JM, Brouqui P, Raoult D. RETRACTED: Hydroxychloroquine and azithromycin as a treatment of COVID-19: results of an open-label non-randomized clinical trial. Int J Antimicrob Agents. 2020 Jul;56(1):105949. doi: 10.1016/j.ijantimicag.2020.105949. Epub 2020 Mar 20. PMID 32205204
- [Background] Cao B, Wang Y, Wen D, Liu W, Wang J, Fan G, Ruan L, Song B, Cai Y, Wei M, Li X, Xia J, Chen N, Xiang J, Yu T, Bai T, Xie X, Zhang L, Li C, Yuan Y, Chen H, Li H, Huang H, Tu S, Gong F, Liu Y, Wei Y, Dong C, Zhou F, Gu X, Xu J, Liu Z, Zhang Y, Li H, Shang L, Wang K, Li K, Zhou X, Dong X, Qu Z, Lu S, Hu X, Ruan S, Luo S, Wu J, Peng L, Cheng F, Pan L, Zou J, Jia C, Wang J, Liu X, Wang S, Wu X, Ge Q, He J, Zhan H, Qiu F, Guo L, Huang C, Jaki T, Hayden FG, Horby PW, Zhang D, Wang C. A Trial of Lopinavir-Ritonavir in Adults Hospitalized with Severe Covid-19. N Engl J Med. 2020 May 7;382(19):1787-1799. doi: 10.1056/NEJMoa2001282. Epub 2020 Mar 18. PMID 32187464
- [Background] Hui DS, Joynt GM, Wong KT, Gomersall CD, Li TS, Antonio G, Ko FW, Chan MC, Chan DP, Tong MW, Rainer TH, Ahuja AT, Cockram CS, Sung JJ. Impact of severe acute respiratory syndrome (SARS) on pulmonary function, functional capacity and quality of life in a cohort of survivors. Thorax. 2005 May;60(5):401-9. doi: 10.1136/thx.2004.030205. PMID 15860716
- [Background] Winters BD, Eberlein M, Leung J, Needham DM, Pronovost PJ, Sevransky JE. Long-term mortality and quality of life in sepsis: a systematic review. Crit Care Med. 2010 May;38(5):1276-83. doi: 10.1097/CCM.0b013e3181d8cc1d. PMID 20308885
- [Background] Rabiee A, Nikayin S, Hashem MD, Huang M, Dinglas VD, Bienvenu OJ, Turnbull AE, Needham DM. Depressive Symptoms After Critical Illness: A Systematic Review and Meta-Analysis. Crit Care Med. 2016 Sep;44(9):1744-53. doi: 10.1097/CCM.0000000000001811. PMID 27153046
- [Background] Semmler A, Widmann CN, Okulla T, Urbach H, Kaiser M, Widman G, Mormann F, Weide J, Fliessbach K, Hoeft A, Jessen F, Putensen C, Heneka MT. Persistent cognitive impairment, hippocampal atrophy and EEG changes in sepsis survivors. J Neurol Neurosurg Psychiatry. 2013 Jan;84(1):62-9. doi: 10.1136/jnnp-2012-302883. Epub 2012 Nov 7. PMID 23134661
- [Background] Mak IW, Chu CM, Pan PC, Yiu MG, Ho SC, Chan VL. Risk factors for chronic post-traumatic stress disorder (PTSD) in SARS survivors. Gen Hosp Psychiatry. 2010 Nov-Dec;32(6):590-8. doi: 10.1016/j.genhosppsych.2010.07.007. Epub 2010 Sep 15. PMID 21112450
- [Background] Rainer TH, Yeung JH, Cheung SK, Yuen YK, Poon WS, Ho HF, Kam CW, Cattermole GN, Chang A, So FL, Graham CA. Assessment of quality of life and functional outcome in patients sustaining moderate and major trauma: a multicentre, prospective cohort study. Injury. 2014 May;45(5):902-9. doi: 10.1016/j.injury.2013.11.006. Epub 2013 Nov 21. PMID 24314871
- [Background] Rainer TH, Hung KKC, Yeung JHH, Cheung SKC, Leung YK, Leung LY, Goggins WB, Ho HF, Kam CW, Cheung NK, Graham CA. Trajectory of functional outcome and health status after moderate-to-major trauma in Hong Kong: A prospective 5 year cohort study. Injury. 2019 May;50(5):1111-1117. doi: 10.1016/j.injury.2019.02.017. Epub 2019 Feb 22. PMID 30827704
- [Background] Rainer TH, Graham CA, Yeung HH, Poon WS, Ho HF, Kam CW, Cameron P. Assessment of long-term functional outcome in patients who sustained moderate or major trauma: a 4-year prospective cohort study. Hong Kong Med J. 2018 Feb;24 Suppl 2(1):30-33. No abstract available. PMID 29938655
- [Background] Lam CL, Tse EY, Gandek B. Is the standard SF-12 health survey valid and equivalent for a Chinese population? Qual Life Res. 2005 Mar;14(2):539-47. doi: 10.1007/s11136-004-0704-3. PMID 15892443
- [Background] Chen J, Wong CK, McGhee SM, Pang PK, Yu WC. A comparison between the EQ-5D and the SF-6D in patients with chronic obstructive pulmonary disease (COPD). PLoS One. 2014 Nov 7;9(11):e112389. doi: 10.1371/journal.pone.0112389. eCollection 2014. PMID 25379673
- [Background] Davis JC, Hsiung GY, Bryan S, Jacova C, Jacova P, Munkacsy M, Cheung W, Lee P, Liu-Ambrose T. Agreement between Patient and Proxy Assessments of Quality of Life among Older Adults with Vascular Cognitive Impairment Using the EQ-5D-3L and ICECAP-O. PLoS One. 2016 Apr 21;11(4):e0153878. doi: 10.1371/journal.pone.0153878. eCollection 2016. PMID 27101402
- See also: World Health Organization. Situation Report-78 HIGHLIGHTS.; 2020 — https://www.who.int/docs/default-source/coronaviruse/situation-reports/20200407-sitrep-78-covid-19.pdf?sfvrsn=bc43e1b_2
- See also: Center for Health Protection G of the HKS. Centre for Health Protection — https://www.chp.gov.hk/en/index.html

DOCUMENTS (2):
  • Informed Consent Form (2020-04-29): https://cdn.clinicaltrials.gov/large-docs/64/NCT04377464/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2020-04-29): https://cdn.clinicaltrials.gov/large-docs/64/NCT04377464/Prot_SAP_001.pdf